CLINICAL TRIAL: NCT05083468
Title: A Randomized, Double-blind, Placebo-controlled, 2-part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of SR750 in Healthy Volunteers
Brief Title: The Safety, Tolerability, and Pharmacokinetics (PK) of SR750 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SR750-101
Record Dates: First submitted 2021-09-27; First posted 2021-10-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SR750 tablet (Experimental): Ascending single and multiple doses of SR750 tablets orally
  Interventions: Drug: SR750 tablet
- matching placebo (Placebo Comparator): Ascending single and multiple doses of matching placebo orally
  Interventions: Drug: matching placebo

INTERVENTIONS:
Drug: SR750 tablet — The volunteers will be orally administrated by single or multiple dose of SR750 tablet with 240 mL water.
  Arms: SR750 tablet
Drug: matching placebo — The volunteers will be orally administrated by single or multiple dose of matching placebo with 240 mL water.
  Arms: matching placebo

SUMMARY:
This study is to evaluate the safety, tolerability, and PK of SR750 in healthy volunteers.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo-controlled, 2-part Phase I study to evaluate the safety, tolerability, and pharmacokinetics of single and multiple ascending doses of SR750 in healthy volunteers. This study includes 2 parts:

Part A is a double-blind, randomized, placebo-controlled, single-dose escalation study of SR750 in healthy volunteers.

Part B is a double-blind, randomized, placebo-controlled, repeated-dose escalation study of SR750 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers will be included in the study if they satisfy all the following criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at Screening.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2, with a body weight ≥ 50 kg for males or ≥ 45 kg for females at screening.
4. Use of tobacco or nicotine-containing products:

   1. Have less than 10 tobacco or nicotine-containing products (including tobacco, e-cigarettes) per week in the last 3 months prior to dosing; abstain from smoking from 7 days prior to dosing until the final follow-up visit;
   2. Have not used any marijuana in the 3 months prior to screening until the end of study.
5. Medically healthy without clinically significant abnormalities at the screening visit, at check-in on Day -1, and pre-dose on Day 1, including:

   1. Physical examination without any clinically relevant findings;
   2. Systolic blood pressure in the range of 90 to 140 mmHg (inclusive) and diastolic blood pressure in the range of 40 to 90 mmHg (inclusive) after 5 minutes in supine position;
   3. Pulse rate in the range of 60 to 100 bpm, inclusive (40-60 bpm [inclusive] may be considered acceptable for athletes or volunteers without clinical significance at the discretion of the PI or designee) after 5 minutes rest in supine position;
   4. Body temperature (tympanic), between 35.5°C and 37.5°C (inclusive);
   5. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests as judged by the Investigator.
6. Conventional 12-lead Electrocardiogram (ECG) recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at the screening visit, on Day 1 and pre-dose on Day 1) consistent with normal cardiac conduction and function, including:

   1. T interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males, and ≤ 470 msec for females;
   2. QRS (wave group of Q, R and S in ECG) duration of ≤ 120 msec;
   3. Electrocardiogram morphology consistent with healthy cardiac ventricular conduction and normal rhythm, and with measurement of the QT interval;
   4. No family history of short or long QT syndrome, or sudden cardiac death;
   5. No history of torsade de pointes or a known arrhythmia.
7. Healthy female volunteers must:

   a) Of non-childbearing potential, defined as: i. Pre-menopausal females with a documented tubal ligation, tubal occlusion procedure followed by a hysterosalpingogram that confirmed bilateral tubal occlusion, bilateral salpingectomy, hysterectomy, bilateral oophorectomy, or other documented medical conditions which cause infertility and are considered to be of non-childbearing potential; Note: "documented" refers to the outcome of the Investigator's/designee's review of the healthy volunteer's medical history for study eligibility, as obtained via a verbal interview with the healthy volunteer or from the healthy volunteer's medical records).

   ii. Postmenopausal, defined as a minimum of 12 months of spontaneous amenorrhea (in questionable cases a blood sample with follicle stimulating hormone [FSH] >40 Million International Units (mIU)/mL is confirmatory).

   b) If of childbearing potential, must have a negative pregnancy test at the screening visit (blood test) and before the first study drug administration (Day -1 urine test). They must agree not to attempt to become pregnant, must not be breastfeeding, must not donate ova from signing the consent form until at least 30 days after the last does of study drug, and must agree to: i. Use 2 forms of highly effective contraceptive method at least 2 weeks prior to screening, between signing consent, during the study, and at least 30 days after the last dose of study therapy, OR ii. Use at least one highly effective contraceptive method, plus an additional barrier-method of contraception at least 2 weeks prior to screening, between signing the consent, during the study, and at least 30 days after the last dose of study drug. Acceptable barrier methods include: female diaphragm condom usage for male partner, OR iii. True abstinence condition at least 2 weeks prior to screening, between signing consent, during the study, and at least 30 days after the last dose of study therapy.

   c) Women of childbearing potential (WOCBP) with solely same sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.
8. Male healthy volunteers, if not surgically sterilised (defined as performed at least 3 months prior to the first dose which could be confirmed by the documentation or verbal interview), must be willing not to donate sperm and, if engaging in sexual intercourse with a female partner who could become pregnant, must be willing to use a condom in addition to having the female partner use a highly effective contraceptive method from signing the consent form until at least 90 days after the last dose of study drug. If engaging in sexual intercourse with a pregnant partner, must be willing to use a barrier-method of contraception. Male healthy volunteers with same-sex partner (abstinence from penile-vaginal intercourse) and male healthy volunteers who are true abstinence are eligible when this is their preferred and usual lifestyle.
9. Male participants must be willing to use a condom if engaging in sexual intercourse with a same sex partner from signing the consent form until study exit.
10. Have suitable venous access for blood sampling.
11. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

Volunteers will be excluded from the study if there is evidence of any of the following:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or significant neurological or psychiatric disease (including history of epilepsy or seizures), including any acute illness or major surgery within the past 3 months determined by the Investigator to be clinically relevant.
2. Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications.
3. Any history of malignant disease in the last 10 years (excludes completely treated cutaneous squamous cell or basal cell carcinoma).
4. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
5. Use of or having plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon, with the exception of topical steroid creams) during the study or within 3 months prior to the first study drug administration.
6. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma glutamyl transferase [GGT]) and bilirubin (total, conjugated and unconjugated) elevated more than 1.2-fold above the upper limit of normal (ULN).
7. Positive test results for active human immunodeficiency virus (HIV-1 and HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
8. Presence or having sequelae of gastrointestinal, liver (including Gilbert's syndrome), kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
9. Estimated creatinine clearance (CrCl) < 80 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN.
10. Regular use of substance abuse or alcohol abuse within 3 months prior to Screening, where "regular" is defined as >21 units of alcohol per week for males and >14 units of alcohol per week for females. One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
11. Positive drug or alcohol test results at the screening visit or at check-in (Day -1) (may be repeated once, if a positive test was recorded in the first instance, at the discretion of the PI or designee).
12. Use of any systemically absorbed prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 × half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol (up to a maximum of 2000 mg per day of paracetamol and per local or national labelling) or hormonal contraceptives.
13. History of demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would increase the risk of having allergic reactions associated with investigational product administration.
14. Known hypersensitivity to any of the study drug ingredients.
15. Use of any vaccinations within 7 days prior to the first study drug administration, or plan to use any vaccinations within 2 weeks after the last dose.
16. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of first study drug administration.
17. The healthy volunteer has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
18. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.
19. Is an employee of an Investigator or Sponsor or an immediate relative of an investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of AEs in healthy volunteers administrated with single and repeated oral doses of SR750 | Up to Day15 for the safety follow up since Day1
  AE: adverse event

OTHER OUTCOMES:
Cmax | Up to Day 10
  Maximum observed concentration
Tmax | Up to Day 10
  Time of peak plasma concentration
Ctrough | Up to Day 10
  Trough concentrations, part B only.
AUC0-t | Up to Day 10
  Area under the concentration-time curve from 0 to time of last quantifiable concentration
AUC0-∞ | Up to Day 10
  Area under the concentration-time curve from 0 to infinity
t1/2 | Up to Day 10
  Apparent terminal elimination half-life
Ae | Up to Day 3, cohort 3 in part A only.
  Cumulative amount of unchanged drug excreted in urine
CLr | Up to Day 3, cohort 3 in part A only.
  Renal clearance

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Johnson, Study Director — Nucleus Network Pty Ltd.
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No